CLINICAL TRIAL: NCT06897891
Title: A Comparative Study on Relieving Postpartum Lumbago with Fire-dragon Cupping Therapy and Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qiaohui Ye (Other)
Responsible Party: Sponsor-Investigator, Qiaohui Ye, Hangzhou Hospital of Traditional Chinese Medicine, Hangzhou Hospital of Traditional Chinese Medicine
Organization: Hangzhou Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023KLL067
Record Dates: First submitted 2025-03-17; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-09

CONDITIONS: Postpartum Low Back Pain; Acupuncture; Core Stability Training; Huolong Tank

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture group (Active Comparator): Acupuncture and moxibustion group combined with core stability training.
  Interventions: Combination Product: Acupuncture combined with core stability training
- Huolong Tank Group (Experimental): Huolong Tank group adopts Huolongcan combined core stability training
  Interventions: Combination Product: Dragon Tank joint core stability training

INTERVENTIONS:
Combination Product: Acupuncture combined with core stability training — All patients were given routine health education guidance and core stability training. Acupuncture group combined with core stability training
  Arms: Acupuncture group
Combination Product: Dragon Tank joint core stability training — All patients were given routine health education guidance and core stability training. Huolong Tank group adopts Huolongcan combined core stability training
  Arms: Huolong Tank Group

SUMMARY:
Abstract: Objective To compare the effects of fire dragon pot therapy and acupuncture on low back pain, lumbar function, self-efficacy and postpartum depression in patients with postpartum low back pain. Methods From April 2024 to September 2024, 84 postpartum patients with low back pain who met the standard of sodium discharge in Hangzhou area were recruited and divided into acupuncture group (routine acupuncture + core stability training (42 cases) and Huolongcan group (42 cases) according to random number table method. Fire dragon pot + core stability training (42 cases), the two groups each intervention 30 min, once every other day, intervention 3 times. Before and after the intervention, the visual Analogue Scale (VAS) was used to evaluate the degree of low back pain, the Oswestry Disability Index (ODI) was used to evaluate the lumbar function, the pain Self-efficacy questionnaire (PSEQ) was used to evaluate the patients' confidence in effectively coping with pain, and the Edinburgh Postpartum Depression Scale (EPDS) was used to evaluate the postpartum depression. The changes of each index before and after intervention were observed.

ELIGIBILITY:
Inclusion Criteria:

* (1) Postpartum 42 days to 1 year; (2) Visual analogue scale (VAS)[7]≥4 points; (3) Have basic reading comprehension ability, be able to fill out questionnaires independently, cooperate with investigation and treatment; (4) Sign informed consent voluntarily.

Exclusion Criteria:

* (1) Tumor, fracture, tuberculosis, bleeding tendency or serious organic disease; (2)Immune system diseases such as ankylosing spondylitis; (3) severe osteoporosis; (4) Patients with Yin deficiency and fire flourishing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
pain score | up to 24 weeks
Lumbar function score | up to 24 weeks
Self-efficacy score | up to 24 weeks
Postpartum depression score | up to 24 weeks

SECONDARY OUTCOMES:
age | baseline, pre-intervention
course of disease | baseline, pre-intervention
  Refers to the total time of disease occurrence, recorded by month.
production mode | baseline, pre-intervention
  It refers to the method that pregnant women choose to give birth, which can be divided into normal birth, caesarean section, and one birth along two births.
parity | baseline, pre-intervention
  It refers to how many times a pregnant woman has been pregnant, including one, two, and three.
Child feeding pattern | baseline, pre-intervention
  Refers to the pregnant women choose to feed the child, including pure breast milk, pure milk powder, breast milk powder mixed feeding
The youngest age | baseline, pre-intervention
body mass index | baseline, pre-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou Hospital of Traditional Chinese Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No